CLINICAL TRIAL: NCT05194644
Title: Effects of Sensorimotor Stimulation Program With and Without Routine Physical Therapy on Balance and Cognitive Performance in Patients With Mild Traumatic Brain Injury: A Randomized Controlled Trial
Brief Title: Sensorimotor Stimulation, Routine Physical Therapy, Balance, Cognitive Performance Mild Traumatic Brain Injury Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Huma Waqar, Effects of sensorimotor stimulation program with and without routine physical therapy on balance and cognitive performance in patients with mild traumatic brain injury: A randomized controlled trial, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/985/2021
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine physical therapy + Sensorimotor stimulation (Experimental): Active and passive Range of motion exercise on upper and lower limb, Transfers from bed to chair, Sit to stand exercise Time duration will be 20 min, Rest period 5 min In Sensory Stimulation Gustatory, Tactile, Olfactory, Visual, Auditory Stimulation will be applied alternatively Time duration will be 4 min In motor stimulation first warm up session for 5-10 min, strengthening exercise, PNF techniques for upper and lower limb, abdominal curls and then different Balance exercises for 6 min 5 times a week
  Interventions: Other: Routine physical therapy+ Sensorimotor stimulation; Other: Routine physical therapy
- Routine physical therapy (Placebo Comparator): Active and passive Range of motion exercise on upper and lower limb, Transfers from bed to chair, Sit to stand exercise Time duration will be 20 min, Rest period 5 min
  Interventions: Other: Routine physical therapy

INTERVENTIONS:
Other: Routine physical therapy+ Sensorimotor stimulation — Gustatory, Tactile, Olfactory, Visual and Auditory Stimulation will be applied in sensory stimulation and in motor stimulation strengthening, Proprioceptive neuromuscular facilitation techniques, Balance exercises will be performed
  Arms: Routine physical therapy + Sensorimotor stimulation
Other: Routine physical therapy — Active and passive Range of motion exercise of upper and lower limb, Transfer from bed to chair, Sit to stand practice

SUMMARY:
Study design: Randomized controlled trial Settings: Physiotherapy department of Allied hospital, Faisalabad Sample size: 27 in each group Control group receive: Routine physical therapy Experimental group receive: Routine physical therapy+ Sensorimotor stimulation

DETAILED DESCRIPTION:
Control group: Routine physical therapy Time duration: 20 min, Rest period: 5 min and treatment will be given 5 days a week and continued for 16 weeks.

Experimental group: Routine physical therapy + Sensorimotor stimulation

Sensorimotor stimulation:

Sensory stimulation:

1. Gustatory stimulation: Irrigation of oral cavity, brushing of teeth and tongue, gum massage, 2ml lemon juice on lateral side of tongue, Time duration will be 4 min.
2. Tactile stimulation: For temperature sensation warm and cold water will applied on different body parts, For touch sensation wet towels and soap will be applied, For pressure sensation body parts will be massaged by lotion, Time duration will be 4 min.
3. Olfactory stimulation: Aromatic stimuli with fragrances to which patient had been familiar e.g. coffee, tea, orange peel and perfume etc. Time duration will be 3 min.
4. Auditory stimulation: Investigator will communicate directly to patients, familiar songs will be utilized, Time duration will be 4 min.
5. Visual stimulation: Colored light, familiar faces, photographs of family members, moving light will be used, Time duration will be 4 min.

Motor stimulation: Warm up session for 5-10 min, Strengthening exercises for upper and lower limb, for trunk flexors and abdominal curls in supine lying, 10rep 2 sets for 3 times a week, Different balance exercise for 6 min 5 times a week.

ELIGIBILITY:
Inclusion Criteria:

* Patient recruit from Outdoor patient department with mild traumatic brain injury having Glasgow coma scale score(13-15)
* Normal intracranial pressure
* Cardiopulmonary stability

Exclusion Criteria:

* Preexisting disabilities
* Suffering from severe medical disease
* Persistent vegetative state
* Patients with opium and drug addicted
* Patients with deafness and delusion disorders

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-07-12 (Estimated); Study Completion 2022-07-22 (Estimated)

PRIMARY OUTCOMES:
Balance | 16th week
  Balance will be measured by Berg balance scale in which (0-20)indicates high fall risk, (21-40) indicates medium fall risk and (41-56) represents low fall risk
Cognitive Performance | 16th week
  Cognitive performance will be measured by Rancho Los Amigos scale that consist of 8 levels. level I indicates no response and needs total assistance whereas level VIII represents purposeful appropriate response and needs stand by assistance,

CONTACTS AND LOCATIONS:
Overall Officials: Huma Waqar, MS PTN*, Principal Investigator — University of Lahore
Locations (1):
- Physiotherapy department of Allied Hospital, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nizamutdinov D, Shapiro LA. Overview of Traumatic Brain Injury: An Immunological Context. Brain Sci. 2017 Jan 23;7(1):11. doi: 10.3390/brainsci7010011. PMID 28124982
- [Background] Capizzi A, Woo J, Verduzco-Gutierrez M. Traumatic Brain Injury: An Overview of Epidemiology, Pathophysiology, and Medical Management. Med Clin North Am. 2020 Mar;104(2):213-238. doi: 10.1016/j.mcna.2019.11.001. PMID 32035565
- [Background] Swanson TM, Isaacson BM, Cyborski CM, French LM, Tsao JW, Pasquina PF. Traumatic Brain Injury Incidence, Clinical Overview, and Policies in the US Military Health System Since 2000. Public Health Rep. 2017 Mar/Apr;132(2):251-259. doi: 10.1177/0033354916687748. Epub 2017 Jan 30. PMID 28135424
- [Background] Finch E, Copley A, Cornwell P, Kelly C. Systematic Review of Behavioral Interventions Targeting Social Communication Difficulties After Traumatic Brain Injury. Arch Phys Med Rehabil. 2016 Aug;97(8):1352-65. doi: 10.1016/j.apmr.2015.11.005. Epub 2015 Dec 8. PMID 26679234